CLINICAL TRIAL: NCT06439511
Title: Comparison of a Non Contact Vital Signs Application (Darwin Edge rVSM) on a Smartphone With Traditional Pulse Oximetry for Heart Rate Measurement: a Prospective Clinical Study
Brief Title: Comparison of a Non Contact Vital Signs Application With Traditional Pulse Oximetry for Heart Rate Measurement
Acronym: Darwin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital du Valais (Other)
Collaborators: University of Lausanne Hospitals (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Darwin
Record Dates: First submitted 2024-05-22; First posted 2024-06-03 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Heart

STUDY DESIGN:
Intervention Model Description: All participants will have heart rate measurement
  1. by pulse oxymetry
  2. by a smartphone application
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulse oxymetry (Active Comparator): Pulse oxymetry is one of the gold standards for non invasive measurement of heart rate.
  Interventions: Device: Pulse oxymetry
- Smartphone app (Experimental): This is a new smartphone application which can potentially measure heart rate in less than 30 seconds.
  Interventions: Device: Darwin smartphone app

INTERVENTIONS:
Device: Darwin smartphone app — The participant must look into the smartphone camera with the Darwin app for about 30 seconds.
  Arms: Smartphone app
Device: Pulse oxymetry — Heart rate will be measured with pulsoe oximetry (gold standard)
  Arms: Pulse oxymetry

SUMMARY:
The investigators want to test the accuracy of the Smartphone application Darwin Edge rVSM in measuring heart rate, as compared to traditional pulsoxymetry. The intervention is to look at the smartphone camera for approximately 30 seconds, and after that to compare the heart rate value with that obtained with a recording by pulsoxymetry.

DETAILED DESCRIPTION:
Participants undergoing a routine perianesthetic consultation at the preanesthetic clinic will be recruited. as a part of routine clinical assessment their heart rate is measured with pulsoxymetry, a non invasive device worn at the fingertip for about 1 minute. this measurement will be compared to the values for heart rate that can be obtaine with the ''Darwin Edge rVSM'' mobile application. this application can be installed on any smartphone. the participant is required to look into the smartphone camera for about 30 seconds. environmental and lighning conditions will be kept stable.

The investigators will do the measurements in 200 participants in order to obtaine values in a population characterized by a variety of phenotypes, in the perioperative setting.

ELIGIBILITY:
Inclusion Criteria:

* Men or women older than 18 years old presenting to the preanesthetic assessment clinic of Valais Hospital
* Subjects that have signed the informed consent form

Exclusion criteria:

* subjects with damaged/injured skin at the face
* Subjects unable to remain still for 30 seconds

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Heart rate | 1 minute
  accuracy of heart rate measurement

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schoettker, MD, Study Director — University of Lausanne Hospitals
Locations (1):
- Valais Hospital, Sion, Valais, Switzerland

IPD SHARING:
Plan to Share IPD: No